CLINICAL TRIAL: NCT07192016
Title: Mechanistic 129-Xe MRI Study of Single Inhaler FF/UMEC/VI Effects in COPD Patients With Persistent, Moderate-severe Dyspnea and/or Poor Health Status With High or Low Risk of Exacerbation
Brief Title: 129-Xe MRI Study of Single Triple Therapy Inhaler Effects in COPD Patients With Moderate-severe Dyspnea and/or Poor Health Status With High or Low Risk of Exacerbation
Acronym: MUST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, Principal Investigator, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROB0054
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Pulmonary Function; COPD; 129-Xenon; Magnetic Resonance Imaging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: single arm, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with persistent moderate-severe COPD (Experimental): Participants with moderate to severe COPD will be evaluated during and after a twelve week trial of triple therapy (ICS/LABA/LAMA) for changes in 129Xe MRI ventilation percent defect, pulmonary function measurements.
  Interventions: Drug: fluticasone furoate(FF)/umeclidinium (UMEC)/vilanterol(VI) (100/62.5/25) mcg

INTERVENTIONS:
Drug: fluticasone furoate(FF)/umeclidinium (UMEC)/vilanterol(VI) (100/62.5/25) mcg — The investigational drug is a single Ellipta inhaler containing 100 ug fluticasone furoate(inhaled corticosteroid), 62.5 ug umeclidinium(long-acting muscarinic antagonist) and 25 ug vilanterol(long-acting β2-adrenergic agonist). The drug is delivered in an Ellipta inhaler in a single dose once daily.
  Other Names: Trelegy

SUMMARY:
The goal of this study is to study how 12-weeks daily (and optional 48-weeks) single inhaler triple therapy (fluticasone furoate (FF)-an inhaled corticosteroid; umeclidinium (UMEC)-a long-acting muscarinic antagonist; vilanterol (VI)-a long-acting β2-adrenergic agonist) works to treat adults with COPD. The investigators will compare the effects of this medication on adults with COPD who are at low risk of a flare-up and adults with COPD who are at high risk of a flare-up. The main questions it aims to answer are:

* Does FF/UMEC/VI improve ventilation defect percent as measured on 129-Xenon MRI in adults with moderate-severe COPD
* Evaluate the relationships between the ventilation defect percent and lung function test results

Participants will:

* Take the inhaler FF/UMEC/VI once daily for 12-weeks (optional 48-weeks)
* visit Robarts 2 times (with optional 3rd visit) for tests and imaging

DETAILED DESCRIPTION:
This study will evaluate 60 COPD patients age 50-85 (equal numbers males and females) with persistent, moderate-severe dyspnea, poor health status and either: 1) low risk of exacerbation (n=30) or moderate-high risk of exacerbation (n=30). Two visits at baseline and 12-weeks are proposed with an optional visit at 48-weeks to assess longitudinal effects of therapy.

At all study visits participants will have vital signs recorded and undergo pre- and post-bronchodilator spirometry, plethysmography, oscillometry, pre-bronchodilator forced exhaled nitric oxide (FeNO) and post-bronchodilator diffusing capacity of the lungs for carbon monoxide (DLco). Participants will undergo pre- and post-bronchodilator 129-Xe MRI and post-bronchodilator chest computed tomography (CT). Participants will complete St. George's Respiratory Questionnaire (SGRQ), Modified Medical Research Council (mMRC), COPD Assessment Test (CAT), Borg rating of perceived exertion questionnaire will be completed before and after the six-minute walk test (6MWT). Participants will have a blood draw for complete blood count (CBC).

ELIGIBILITY:
Inclusion Criteria:

* patient understands study procedures and is willing to participate in the study as indicated by the patient's signature
* provision of written, informed consent prior to any study specific procedures
* males and females 50-85 years of age
* stable COPD, currently on dual therapy LAMA/LABA or ICS/LABA or initial maintenance therapy for at least 3 months
* mMRC score ≥2 and/or CAT score ≥10
* Low risk subgroup: participant has experienced ≤1 exacerbation in the past year and no hospitalizations for COPD High risk subgroup: participant has experienced ≥2 exacerbations in the past year
* Female of childbearing potential (after menarche) must ensure that they are using an effective form of birth control for at least 2 months prior to each imaging visit. Examples of effective birth control include:

  1. True sexual abstinence
  2. A vasectomized sexual partner
  3. Implanon®
  4. Female sterilization by tubal occlusion
  5. Effective intrauterine device (IUD)/levonogestrel intrauterine system (IUS)
  6. Depo-Provera™ injections
  7. Oral contraceptive
  8. Evra Patch™
  9. Nuvaring™
* Female permanently sterile due to: 1) documented hysterectomy, 2) documented bilateral salpingectomy, and 3) documented bilateral oophorectomy
* Postmenopausal female: defined as female with no menses for 12 months without an alternative medical cause
* Females of childbearing potential (after menarche) must agree to use a highly effective form of birth control, as defined above, from enrollment, throughout the study duration, and 8 weeks after last dose of study drug, with negative urine pregnancy test taken within 24 hr of any planned CT examination at Visit-1 through Visit 3
* Male participants who are sexually active with a woman who can still have children, must agree to use a double barrier method of contraception (male condom with diaphragm or male condom with cervical cap) from the first dose of the study drug until 8 weeks after last dose

Exclusion Criteria:

* Patient has an implanted mechanically, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist)
* In the investigator's opinion, participant suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI or CT, such as severe claustrophobia
* Participants who are pregnant, breastfeeding or have a positive pregnancy test at initial screening visit
* Participant is unable to perform spirometry or plethysmography maneuvers
* Participant is unable to perform MRI and CT breath-hold maneuvers
* Participant has an unstable cardiovascular, gastro-intestinal, hepatic, renal, neurologic, metabolic or psychiatric disease
* Participation in any clinical trial of an investigational agent or procedure within three months prior to screening or during the study
* Known history of allergy or reaction to the study drug formulation
* Participant has a blood pressure of >150 mmHg systolic or >95 mmHg diastolic on more than 2 measurements done >5 minutes apart at Visit-1
* Participants with a recently (<2 months) documented diagnosis of asthma

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Measure the effect of FF/UMEC/VI therapy on VDP | 12-weeks and optional 48-weeks
  Measured using 129-xenon MRI ventilation defect percent
Measure the effect of FF/UMEC/VI on FEV1 | at 12-weeks and optional 48-weeks
  Measured by the forced expiratory volume at 1 second

SECONDARY OUTCOMES:
Evaluate the relationship between MRI VDP and lung function | 12-weeks and optional 48-weeks
  measured using MRI ventilation defect percent and forced expiratory volume at 1 second
Evaluate the relationship between MRI VDP and SGRQ score | 12-weeks and optional 48-weeks
  measured using 129-xenon MRI ventilation defect percent and St. George's Respiratory Questionnaire score
Evaluate the relationship between MRI VDP and CAT score | 12-weeks and optional 48-weeks
  Measured using 129-xenon MRI ventilation defect percent and COPD Assessment Test score
Evaluate the relationship between MRI VDP and mMRC score | 12-weeks and optional 48-weeks
  Measured using 129-xenon MRI ventilation defect percent and modified Medical Research Council questionnaire score
Evaluate the relationship between MRI VDP and 6MWD | 12-weeks and optional 48-weeks
  Measured using 129-xenon MRI ventilation defect percent and six-minute walk distance.
Evaluate and compare potential differences in MRI VDP response among patients with low- and high-risk of exacerbation. | 12-weeks and optional 48-weeks
  Measured using 129-xenon MRI ventilation defect percent and comparing exacerbation rates across patients with low- and high-risk of exacerbation.
Evaluate the relationship between MRI VDP and blood inflammatory markers | 12-weeks and optional 48-weeks
  Measured using 129-xenon MRI ventilation defect percent and blood eosinophil count
Evaluate the relationship between MRI VDP and CT measurements | 12-weeks and optional 48-weeks
  Measured using 129-xenon MRI ventilation defect percent and CT mucus-score
Evaluate change in VDP as a predictor of annualized exacerbation rate | 12-weeks and optional 48-weeks
  Measured using change in 129-xenon MRI ventilation defect percent with annualized exacerbation rate as reported by the participant
Evaluate the relationship between MRI VDP and lung volume | 12-weeks and optional 48-weeks
  Measured using MRI ventilation defect percent and forced vital capacity
Evaluate the relationship between MRI VDP and CT measurements | 12-weeks and optional 48-weeks
  Measured using MRI ventilation defect percent and CT mucus-count
Evaluate the relationship between MRI VDP and CT measurements | 12-weeks and optional 48-weeks
  Measured using MRI ventilation defect percent and CT mucus-volume

CONTACTS AND LOCATIONS:
Overall Officials: Grace Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGavin CR, Artvinli M, Naoe H, McHardy GJ. Dyspnoea, disability, and distance walked: comparison of estimates of exercise performance in respiratory disease. Br Med J. 1978 Jul 22;2(6132):241-3. doi: 10.1136/bmj.2.6132.241. PMID 678885
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Kaushik SS, Robertson SH, Freeman MS, He M, Kelly KT, Roos JE, Rackley CR, Foster WM, McAdams HP, Driehuys B. Single-breath clinical imaging of hyperpolarized (129)Xe in the airspaces, barrier, and red blood cells using an interleaved 3D radial 1-point Dixon acquisition. Magn Reson Med. 2016 Apr;75(4):1434-43. doi: 10.1002/mrm.25675. Epub 2015 May 18. PMID 25980630
- [Background] Costella S, Kirby M, Maksym GN, McCormack DG, Paterson NA, Parraga G. Regional pulmonary response to a methacholine challenge using hyperpolarized (3)He magnetic resonance imaging. Respirology. 2012 Nov;17(8):1237-46. doi: 10.1111/j.1440-1843.2012.02250.x. PMID 22889229
- [Background] Kirby M, Heydarian M, Svenningsen S, Wheatley A, McCormack DG, Etemad-Rezai R, Parraga G. Hyperpolarized 3He magnetic resonance functional imaging semiautomated segmentation. Acad Radiol. 2012 Feb;19(2):141-52. doi: 10.1016/j.acra.2011.10.007. Epub 2011 Nov 21. PMID 22104288
- [Background] King GG, Bates J, Berger KI, Calverley P, de Melo PL, Dellaca RL, Farre R, Hall GL, Ioan I, Irvin CG, Kaczka DW, Kaminsky DA, Kurosawa H, Lombardi E, Maksym GN, Marchal F, Oppenheimer BW, Simpson SJ, Thamrin C, van den Berge M, Oostveen E. Technical standards for respiratory oscillometry. Eur Respir J. 2020 Feb 27;55(2):1900753. doi: 10.1183/13993003.00753-2019. Print 2020 Feb. PMID 31772002
- [Background] Bhakta NR, McGowan A, Ramsey KA, Borg B, Kivastik J, Knight SL, Sylvester K, Burgos F, Swenson ER, McCarthy K, Cooper BG, Garcia-Rio F, Skloot G, McCormack M, Mottram C, Irvin CG, Steenbruggen I, Coates AL, Kaminsky DA. European Respiratory Society/American Thoracic Society technical statement: standardisation of the measurement of lung volumes, 2023 update. Eur Respir J. 2023 Oct 12;62(4):2201519. doi: 10.1183/13993003.01519-2022. Print 2023 Oct. PMID 37500112
- [Background] Graham BL, Brusasco V, Burgos F, Cooper BG, Jensen R, Kendrick A, MacIntyre NR, Thompson BR, Wanger J. 2017 ERS/ATS standards for single-breath carbon monoxide uptake in the lung. Eur Respir J. 2017 Jan 3;49(1):1600016. doi: 10.1183/13993003.00016-2016. Print 2017 Jan. PMID 28049168
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Schmidt MH, Marshall J, Downie J, Hadskis MR. Pediatric magnetic resonance research and the minimal-risk standard. IRB. 2011 Sep-Oct;33(5):1-6. No abstract available. PMID 22043743
- [Background] Shukla Y, Wheatley A, Kirby M, Svenningsen S, Farag A, Santyr GE, Paterson NA, McCormack DG, Parraga G. Hyperpolarized 129Xe magnetic resonance imaging: tolerability in healthy volunteers and subjects with pulmonary disease. Acad Radiol. 2012 Aug;19(8):941-51. doi: 10.1016/j.acra.2012.03.018. Epub 2012 May 15. PMID 22591724
- [Background] Driehuys B, Martinez-Jimenez S, Cleveland ZI, Metz GM, Beaver DM, Nouls JC, Kaushik SS, Firszt R, Willis C, Kelly KT, Wolber J, Kraft M, McAdams HP. Chronic obstructive pulmonary disease: safety and tolerability of hyperpolarized 129Xe MR imaging in healthy volunteers and patients. Radiology. 2012 Jan;262(1):279-89. doi: 10.1148/radiol.11102172. Epub 2011 Nov 4. PMID 22056683
- [Background] Kirby M, Pike D, Sin DD, Coxson HO, McCormack DG, Parraga G. COPD: Do Imaging Measurements of Emphysema and Airway Disease Explain Symptoms and Exercise Capacity? Radiology. 2015 Dec;277(3):872-80. doi: 10.1148/radiol.2015150037. Epub 2015 Jul 7. PMID 26151081
- [Background] Kirby M, Eddy RL, Pike D, Svenningsen S, Coxson HO, Sin DD, McCormack DG, Parraga G; Canadian Respiratory Research Network. MRI ventilation abnormalities predict quality-of-life and lung function changes in mild-to-moderate COPD: longitudinal TINCan study. Thorax. 2017 May;72(5):475-477. doi: 10.1136/thoraxjnl-2016-209770. Epub 2017 Mar 3. PMID 28258250
- [Background] Kirby M, Kanhere N, Etemad-Rezai R, McCormack DG, Parraga G. Hyperpolarized helium-3 magnetic resonance imaging of chronic obstructive pulmonary disease exacerbation. J Magn Reson Imaging. 2013 May;37(5):1223-7. doi: 10.1002/jmri.23896. Epub 2012 Nov 2. PMID 23124806
- [Background] Kirby M, Svenningsen S, Kanhere N, Owrangi A, Wheatley A, Coxson HO, Santyr GE, Paterson NA, McCormack DG, Parraga G. Pulmonary ventilation visualized using hyperpolarized helium-3 and xenon-129 magnetic resonance imaging: differences in COPD and relationship to emphysema. J Appl Physiol (1985). 2013 Mar 15;114(6):707-15. doi: 10.1152/japplphysiol.01206.2012. Epub 2012 Dec 13. PMID 23239874
- [Background] Kirby M, Mathew L, Wheatley A, Santyr GE, McCormack DG, Parraga G. Chronic obstructive pulmonary disease: longitudinal hyperpolarized (3)He MR imaging. Radiology. 2010 Jul;256(1):280-9. doi: 10.1148/radiol.10091937. PMID 20574101